CLINICAL TRIAL: NCT06474936
Title: Nutritional Health Assistance for Adapting Food Culture to the Mediterranean Pattern for International Students at the University of Pavia (MeditEat)
Brief Title: Adapting Food Culture to the Mediterranean Pattern for International Students in Italy
Acronym: MeditEat
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24013/2024
Record Dates: First submitted 2024-06-13; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Physical Inactivity; Eating Disorders; Eating Habit; Diet, Healthy; Diet Habit
MeSH Terms: conditions — Sedentary Behavior; Feeding and Eating Disorders; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Food habits education regarding the Mediterranean diet adapted according to the country of origin.
  Interventions: Behavioral: Food education

INTERVENTIONS:
Behavioral: Food education — During the consultations are planned at least 6 nutritional education sessions in which the general nutritional advice provided by the Mediterranean Diet will be exposed, and some paper materials can be delivered according to the needs of each individual. 3 in-person meetings and 3 online meetings are planned. Both online and in-person food education sessions will be conducted by experienced nutrition experts monthly. These sessions will cover a range of topics, including the principles of the Mediterranean diet, practical cooking skills, meal-planning strategies, and tips for incorporating Mediterranean-style dishes into daily life
  Other Names: Nutritional education

SUMMARY:
The goal of this clinical trial is to describe the adherence to the Mediterranean diet, the nutritional status, the level of physical activity, and possible eating disorders in international students attending the University of Pavia before and after a food education intervention. The main questions it aims to answer are:

Does the intervention of food education change the nutritional status of the international students of the University of Pavia? Does the intervention of food education change the level of physical activity of international students of the University of Pavia? Does the intervention of food education change the possible risk of eating disorders related to the possible change of diet from the country of origin of international students? Researchers will compare the measurements done at the first meeting to the measurements made at the last meeting (6 months) to see if the food educational intervention helped the students.

Participants will:

* have the body composition analysed by anthropometric measurements (weight, height, electric bio impedance)
* Receive personalized guidance and support from our team of experts for 6 months.

Visit the clinic 3 times (beginning, 3 months, and by the end of 6 months) for check-ups and tests, and participate in online meetings the other 3 months (second, fourth, and fifth).

Answer online questionnaires and perform a 3-day food diary (beginning, 3 months, and by the end of 6 months).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Able to understand English or Italian
* Nationality diverse than Italian
* Absence of major morbidities that interfere with food choices, such as diabetes, hypertension, renal dysfunction, etc.

Exclusion Criteria:

* ≤18 years old;
* Italian nationality;
* Presence of major morbidities that interfere with food choices, such as diabetes, hypertension, renal dysfunction, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Mediterranean Diet Adhrence | 6 months
  Mediterranean Diet Score9 (MEDI-LITE): a tool for measuring adherence to the Mediterranean diet. It assigns points based on the frequency of consumption of nine food categories: (1) fruit; (2) vegetables; (3) cereal grains; (4) legumes; (5) fish and fish products; (6) meat and meat products; (7) dairy products; (8) alcohol intake and (9) olive oil. The final score was obtained by summing these values, and it varies from 0 (low adherence) to 18 (high adherence).

SECONDARY OUTCOMES:
Short Form Health Survey | 6 months
  The SF-36, short for the 36-Item Short Form Health Survey, is a widely used and well-established tool in the field of health-related quality of life assessment. Higher scores mean a better outcome.
Weight | 6 months
  Standardised measurements: weight in kilograms
Dietary evaluation | 6 months
  Food diaries: will be requested for all participants a 3-day food diary by baseline, 3 and 6 months. These diaries will be calculated by macro and micronutrient intake. Food frequency questionnaire 110 items will be applied at T0, T3 and T6. The presence of typical Mediterranean food will be considered as a marker of acculturation.
Height | 6 months
  Standardised measurements: Height in centimeters (cm)
Skin folds | 6 months
  Skin folds (in millimeters) will be recorded by an expert dietician according to standardized procedures (Lohman, 1988).
Body Composition BIA | 6 months
  The Bioelectrical Impedance Analysis, which is a non-invasive and commonly used method for assessing body composition (BIA 101 BIVA PROTM- AKERN) in terms of percentage of fat mass (%).
Physical activity | 6 months
  Standardized tool used to assess an individual's physical activity levels and patterns. Higher scores mean a better outcome.
Fat mass | 6 months
  The evaluation of body composition will be carried out on the basis of skinfold measurements, and using the Bioelectrical Impedance Analysi. The median from the 2 measurements (skinfold and BIA) for fat mass will be used (in percentage).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Laboratory of Food Education and Sport Nutrition, Department of Public Health, Experimental and Forensic Medicine, Pavia
  - University of Pavia, Pavia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neri LCL, Fiorini S, Bosio F, Guglielmetti M, Ferraro OE, Tagliabue A, Ferraris C. Nutritional health assistance for adapting food culture to the Mediterranean pattern for international students: study protocol. Int J Food Sci Nutr. 2025 Nov;76(7):725-735. doi: 10.1080/09637486.2025.2561711. Epub 2025 Sep 25. PMID 40995823